CLINICAL TRIAL: NCT04967716
Title: Genetics of Charcot-Marie-Tooth Dystrophy and Related Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018206
Record Dates: First submitted 2021-06-27; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Peroneal Muscular Atrophy
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peroneal muscular atrophy: Peroneal muscular atrophy (Charcot-Marie-Tooth, CMT) is a group of genetic diseases that invade the peripheral nervous system with very high genetic heterogeneity. It was proposed by Charcot, Marie of France and Tooth of the United Kingdom in 1886. The prevalence is about 1/2500-4000. It is the most common hereditary peripheral neuropathy. Inheritance includes all forms of Mendelian inheritance. The typical clinical manifestations are progressive, length-dependent limb weakness and atrophy, accompanied by hypoesthesia and weakened tendon reflexes.
  Interventions: Other: basic information; Other: venous blood test

INTERVENTIONS:
Other: basic information — Demographic data registration, medical history inquiry, physical examination; electromyography, nerve conduction velocity examination; CMT nerve function score;
Other: venous blood test — The specific method is as follows: 12ml of peripheral blood is drawn from the peripheral vein, and EDTA is used for anticoagulation. No fasting is required before blood draw, and there is no time limit. Part of the specimens submitted for inspection are sent to a qualified genetic testing company for examination, and the fees are charged in accordance with the corresponding charging standards set by the hospital. The remaining part of the sample will be stored or accumulated for a period of time, and the DNA will be extracted and stored in the sample library.

SUMMARY:
This is a cross-sectional study to clarify the gene lineage distribution of CMT genes in CMT patients in my country, draw a frequency map of CMT gene distribution, and assist in determining the genetic diagnosis strategy of CMT diseases. All patients will be collected for clinical and electrophysiological data. Patients and families who meet the enrollment criteria will be tested for blood tests.

DETAILED DESCRIPTION:
[Background] Peroneal muscular atrophy (Charcot-Marie-Tooth, CMT) is a group of the most common hereditary peripheral neuropathy, with a prevalence of about 1/2500-4000. The inheritance mode can be autosomal dominant inheritance, autosomal recessive inheritance, X-linked dominant inheritance and X-linked recessive inheritance. The typical clinical manifestations are progressive, length-dependent weakness and atrophy of the distal limbs, accompanied by hypoesthesia and weakened tendon reflexes. But the generalized peroneal muscular atrophy also includes hereditary motor neuropathy and hereditary sensory neuropathy, which represents the evolution of a disease spectrum from motor nerve to motor sensory nerve and sensory nerve, collectively referred to as CMT and its related diseases. CMT can be divided into demyelinating type (CMT1), axonal type (CMT2) and intermediate type. There are more than 80 kinds of genes discovered so far, and genetic diagnosis plays a vital role in the treatment of peroneal muscular atrophy and genetic counseling.

[Purpose]

1. To clarify the gene lineage distribution of CMT genes in CMT patients in my country, draw a frequency map of CMT gene distribution, and assist in determining the genetic diagnosis strategy of CMT diseases;
2. Discover new mutations and newly published types of known genes, and perform gene-phenotype correlation analysis
3. Perform whole-exome sequencing on some families that have not been clearly diagnosed to find new pathogenic genes or related genes of CMT, so as to enrich the genetic and clinical types of CMT.

[Design] This is a cross-sectional study. All patients will be collected for clinical and electrophysiological data. Patients and families who meet the enrollment criteria will be tested for blood tests. The inspection strategies are as follows: (1) Use MLPA method for PMP22 gene Duplicate or deletion mutation check (charge); (2)) Use high-throughput sequencing method to detect the currently known gene panel (gene panel) (charge); (3) Check the process (1) and (2) Some patients and families whose disease-causing genes have not been detected by the inspection methods are tested by whole-exome sequencing (scientific research, free of charge).

ELIGIBILITY:
Inclusion Criteria:

* Meet the clinical diagnostic criteria of peroneal muscular atrophy; Sign informed consent

Exclusion Criteria:

* Those who have recently received blood transfusion treatment will not be able to collect blood samples.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Peroneal muscular atrophy is a group of genetic diseases with very high genetic heterogeneity that violates the peripheral nervous system. The typical clinical manifestations are progressive, length-dependent limb weakness and atrophy, accompanied by hypoesthesia and weakened tendon reflexes.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
allele frequency of CMT genes | 1 month
  Observed values of allele frequency of CMT genes
genotype frequency of CMT genes | 1 month
  Observed values genotype frequency of CMT genes

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxuan Liu, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No